CLINICAL TRIAL: NCT02390609
Title: Open-Label, Randomized, Parallel Group, 3- or 4-Way Crossover Bioavailability Study of Ibrutinib Suspension and Sprinkle Formulations Compared to Capsules in Healthy Adults
Brief Title: A Crossover Study to Evaluate the Bioavailability of Ibrutinib Suspension and Sprinkle Formulations Compared to Capsules in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR106946; 2015-000155-25 (EudraCT Number); PCI-32765CLL1015 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Healthy; Ibrutinib; Bioavailability
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Group 1: Sequence 1 (ABC) (Experimental): Participants will receive Treatment A (Ibrutinib 560 milligram [mg] capsules [reference] under fasted conditions) in Period 1; followed by Treatment B (Ibrutinib 560 mg suspension under fasted conditions) in Period 2; followed by Treatment C (Ibrutinib 560 mg suspension under fed conditions) in Period 3. A washout period of 7 (plus [+] / minus [-] 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment B); Drug: Ibrutinib (Treatment C)
- Group 1: Sequence 2 (BCA) (Experimental): Participants will receive Treatment B (Ibrutinib 560 mg suspension under fasted conditions) in Period 1; followed by Treatment C (Ibrutinib 560 mg suspension under fed conditions) in Period 2; followed by Treatment A (Ibrutinib 560 mg capsules [reference] under fasted conditions) in Period 3. A washout period of 7 (+/- 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment B); Drug: Ibrutinib (Treatment C)
- Group 1: Sequence 3 (CAB) (Experimental): Participants will receive Treatment C (Ibrutinib 560 mg suspension under fed conditions) in Period 1; followed by Treatment A (Ibrutinib 560 mg capsules [reference] under fasted conditions) in Period 2; followed by Treatment B (Ibrutinib 560 mg suspension under fasted conditions) in Period 3. A washout period of 7 (+/- 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment B); Drug: Ibrutinib (Treatment C)
- Group 1: Sequence 4 (ACB) (Experimental): Participants will receive Treatment A (Ibrutinib 560 mg capsules [reference] under fasted conditions) in Period 1; followed by Treatment C (Ibrutinib 560 mg suspension under fed conditions) in Period 2; followed by Treatment B (Ibrutinib 560 mg suspension under fasted conditions) in Period 3. A washout period of 7 (+/- 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment B); Drug: Ibrutinib (Treatment C)
- Group 1: Sequence 5 (BAC) (Experimental): Participants will receive Treatment B (Ibrutinib 560 mg suspension under fasted conditions) in Period 1; followed by Treatment A (Ibrutinib 560 mg capsules [reference] under fasted conditions) in Period 2; followed by Treatment C (Ibrutinib 560 mg suspension under fed conditions) in Period 3. A washout period of 7 (+/- 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment B); Drug: Ibrutinib (Treatment C)
- Group 1: Sequence 6 (CBA) (Experimental): Participants will receive Treatment C (Ibrutinib 560 mg suspension under fed conditions) in Period 1; followed by Treatment B (Ibrutinib 560 mg suspension under fasted conditions) in Period 2; followed by Treatment A (Ibrutinib 560 mg capsules [reference] under fasted conditions) in Period 3. A washout period of 7 (+/- 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment B); Drug: Ibrutinib (Treatment C)
- Group 2: Sequence 1 (AFDE) (Experimental): Participants will receive Treatment A (Ibrutinib 560 mg capsules [reference] under fasted conditions) in Period 1; followed by Treatment F (Ibrutinib 560 mg sprinkle capsule granules suspended in water under fasted conditions) in Period 2; followed by Treatment D (Ibrutinib 560 mg sprinkle capsule granules under fasted conditions) in Period 3; followed by Treatment E (Ibrutinib 560 mg sprinkle capsule granules under fed conditions) in Period 4. A washout period of 7 (+/- 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment D); Drug: Ibrutinib (Treatment E); Drug: Ibrutinib (Treatment F)
- Group 2: Sequence 2 (DAEF) (Experimental): Participants will receive Treatment D (Ibrutinib 560 mg sprinkle capsule granules under fasted conditions) in Period 1; followed by Treatment A (Ibrutinib 560 mg capsules [reference] under fasted conditions) in Period 2; followed by Treatment E (Ibrutinib 560 mg sprinkle capsule granules under fed conditions) in Period 3; followed by Treatment F (Ibrutinib 560 mg sprinkle capsule granules suspended in water under fasted conditions) in Period 4. A washout period of 7 (+/- 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment D); Drug: Ibrutinib (Treatment E); Drug: Ibrutinib (Treatment F)
- Group 2: Sequence 3 (EDFA) (Experimental): Participants will receive Treatment E (Ibrutinib 560 mg sprinkle capsule granules under fed conditions) in Period 1; followed by Treatment D (Ibrutinib 560 mg sprinkle capsule granules under fasted conditions) in Period 2; followed by Treatment F (Ibrutinib 560 mg sprinkle capsule granules suspended in water under fasted conditions) in Period 3; followed by Treatment A (Ibrutinib 560 mg capsules [reference] under fasted conditions) in Period 4. A washout period of 7 (+/- 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment D); Drug: Ibrutinib (Treatment E); Drug: Ibrutinib (Treatment F)
- Group 2: Sequence 4 (FEAD) (Experimental): Participants will receive Treatment F (Ibrutinib 560 mg sprinkle capsule granules suspended in water under fasted conditions) in Period 1; followed by Treatment E (Ibrutinib 560 mg sprinkle capsule granules under fed conditions) in Period 2; followed by Treatment A (Ibrutinib 560 mg capsules [reference] under fasted conditions) in Period 3; followed by Treatment D (Ibrutinib 560 mg sprinkle capsule granules under fasted conditions) in Period 4. A washout period of 7 (+/- 2) days will be maintained between each treatment period.
  Interventions: Drug: Ibrutinib (Treatment A) [Reference]; Drug: Ibrutinib (Treatment D); Drug: Ibrutinib (Treatment E); Drug: Ibrutinib (Treatment F)

INTERVENTIONS:
Drug: Ibrutinib (Treatment A) [Reference] — Participants will receive Ibrutinib 560 milligram (mg) (4*140 mg) capsule as Treatment A under fasted conditions in one of the treatment periods.
Drug: Ibrutinib (Treatment B) — Participants will receive Ibrutinib 560 mg suspension as Treatment B under fasted conditions in one of the treatment periods.
  Arms: Group 1: Sequence 1 (ABC); Group 1: Sequence 2 (BCA); Group 1: Sequence 3 (CAB); Group 1: Sequence 4 (ACB); Group 1: Sequence 5 (BAC); Group 1: Sequence 6 (CBA)
Drug: Ibrutinib (Treatment C) — Participants will receive Ibrutinib 560 mg suspension as Treatment C under fed (high-fat) conditions in one of the treatment periods.
  Arms: Group 1: Sequence 1 (ABC); Group 1: Sequence 2 (BCA); Group 1: Sequence 3 (CAB); Group 1: Sequence 4 (ACB); Group 1: Sequence 5 (BAC); Group 1: Sequence 6 (CBA)
Drug: Ibrutinib (Treatment D) — Participants will receive Ibrutinib 560 mg sprinkle capsule granules as Treatment D under fasted conditions in one of the treatment periods.
  Arms: Group 2: Sequence 1 (AFDE); Group 2: Sequence 2 (DAEF); Group 2: Sequence 3 (EDFA); Group 2: Sequence 4 (FEAD)
Drug: Ibrutinib (Treatment E) — Participants will receive Ibrutinib 560 mg sprinkle capsule granules as Treatment E under fed (high-fat) conditions in one of the treatment periods.
  Arms: Group 2: Sequence 1 (AFDE); Group 2: Sequence 2 (DAEF); Group 2: Sequence 3 (EDFA); Group 2: Sequence 4 (FEAD)
Drug: Ibrutinib (Treatment F) — Participants will receive Ibrutinib 560 mg sprinkle capsule granules suspended in water as Treatment F under fasted conditions in one of the treatment periods.
  Arms: Group 2: Sequence 1 (AFDE); Group 2: Sequence 2 (DAEF); Group 2: Sequence 3 (EDFA); Group 2: Sequence 4 (FEAD)

SUMMARY:
The purpose of this study is to assess the relative bioavailability (the extent to which a drug or other substance becomes available to the body) of ibrutinib in healthy adults following single oral dose administration of suspension and sprinkle formulations under fed and fasted conditions compared with capsules under fasted conditions.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (study medication assigned to participants by chance), 3- or 4-way crossover (participants may receive different interventions sequentially during the trial), and single-center study of ibrutinib. The duration of study will be approximately 67 to 83 days per participant. The study consists of 3 parts: Screening (28 days before study commences on Day 1); Open-label Treatment (consists of 6 treatments, either Ibrutinib capsule or suspension or sprinkle capsule granules under fed or fasted condition), in subsequent 3 periods for Group 1 and 4 periods for Group 2, each separated with washout period of 7 (plus [+] / minus [-] 2) days; and follow up Phase (up to 10 + / - 2 days after last study drug administration). All the eligible participants will be randomly assigned to 1 of the 6 (Group 1) or 4 (Group 2) treatment sequences. In fasted conditions, study drug will be administered following a 10-hour overnight fast. In fed conditions, participants will also fast from food for 10 hours, but will consume a high fat breakfast within a 30-minute period. Study drug will be administered 2 hours after the breakfast. Participants will not be allowed to have food until 4 hours of drug administration. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Relative bioavailability of Ibrutinib will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* If a woman, must not be of childbearing potential: postmenopausal ( greater than [>] 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) >40 International units [IU]/ Liter [L]); surgically sterile
* If a woman, must have a negative serum β-human chorionic gonadotropin (hCG) pregnancy test at Screening and a negative urine pregnancy test on Day-1 of the each treatment period
* If a man who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (eg, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index (BMI; weight [kg]/height^2 [m]^2) between 18 and 30 Kilogram (kg)/ meter^2 (m^2) (inclusive), and body weight not less than 50 kg

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (creatinine clearance below 60 milliliter [mL]/ minute [min]), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, coagulation, clinical chemistry, at Screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at Screening as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled until completion of the study
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) (DSM-IV) criteria within 2 years before Screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) at Screening and Day-1 of the each treatment period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Ibrutinib | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The Cmax is the maximum observed plasma concentration of Ibrutinib.
Time to Reach the Maximum Plasma Concentration (Tmax) of Ibrutinib | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The Tmax is the time to reach the maximum observed plasma concentration of Ibrutinib.
Area Under the Plasma Concentration-Time Curve From 0 to 24 Hours (AUC[0-24]) Post Dose of Ibrutinib | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The AUC (0-24hrs) is the area under the plasma Ibrutinib concentration-time curve from 0 to 24 hours post dosing.
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Observed Quantifiable Concentration (AUC [0-last]) of Ibrutinib | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The AUC (0-last) is the area under the plasma Ibrutinib concentration-time curve from time 0 to time of the last observed quantifiable concentration (C[last]).
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of Ibrutinib | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The AUC (0-infinity) is the area under the plasma Ibrutinib concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma Ibrutinib concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Percentage of Area Under the Plasma Concentration-Time Curve Obtained by Extrapolation (%AUC[infinity,ex]) | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The %AUC(infinity,ex) is calculated by dividing the difference of AUC(0-infinity) and AUC(0-last) by AUC(0-infinity) and then multiplying by 100, (AUC[0-infinity] - AUC[0-last])*100/AUC[0-infinity].
Terminal Half-life (t[1/2]) of Ibrutinib | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The t(1/2) is defined as 0.693/Lambda (z).
Elimination Rate Constant (Lambda [z]) of Ibrutinib | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The Lambda (z) determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve.
Adjusted Coefficient of Determination (r^2 [adjusted]) | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The r^2 [adjusted] for the number of points used in the estimation of lambda[z].
Relative Bioavailability (Frel) of Ibrutinib | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  The Frel will be calculated as individual Cmax and AUC treatment ratios (for the comparison of food effect). Calculated as: [(AUC[0-infinity][test]/AUC[0-infinity][ref])*(Dose[ref]/Dose[test])]*100.
Metabolite to Parent Ratio for Maximum Plasma Concentration (Cmax) of Ibrutinib | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 1 of each period
  Metabolite to parent drug ratio for maximum observed plasma concentration of Ibrutinib.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (10 plus [+] / minus [-] 2 days after last dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development Clinical Trial, Study Director — Janssen Research & Development
Locations (1):
- Antwerp, Belgium